CLINICAL TRIAL: NCT01325155
Title: Effect of Air Pollution in the Haifa Bay Area on Cardiovascular Morbidity and Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Haim Hammerman Chief of Cardiology, Rambam Medical Center
Other Study IDs: 0043-11CTIL
Record Dates: First submitted 2011-03-27; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Acute Coronary Syndrome; Heart Failure; Arrhythmia
Keywords: Air Pollution; particulate matter; cardiovascular Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The association between exposure to ambient air pollution and pulmonary disease has been well established.To date no study has assessed the burden of cardiovascular disease in Israel and its relation to ambient air pollution.

The Haifa Bay Area has a long history of industrialization including possessing the nation's largest oil refineries, oil-fired power plant, agrochemical and cement producers, industrial incinerators and the Eastern Mediterranean's busiest port. The presence of industrial and mobile sources, combined with a basin effect has contributed to air pollution in the Haifa Bay Area and has raised concerns about potential health effects.

Research Objectives

* Determine if the increased rate of cardiovascular mortality in Haifa is associated with PM 2.5 concentrations.
* Assess effect modification in diverse sub-populations.
* If an association does exist, assess the economic burden of PM 2.5 associated cardiovascular morbidity and mortality.
* Design prediction models of daily cardiovascular emergency department visits based on daily and seasonal variation of air pollution.

DETAILED DESCRIPTION:
The association between exposure to ambient air pollution and pulmonary disease has been well established. Recent studies have attempted to investigate the effect of air pollution, specifically exposure to PM 2.5, on cardiovascular outcomes. Acute exposure to PM 2.5 is associated with increased heart rate, decreased heart rate variability, and increased incidence of cardiac arrhythmia. Population based research from the United States and Europe has demonstrated increased rates of emergency room visits, hospitalization and cardiovascular morbidity in association with increased daily concentrations of fine particulates.

To date no study has looked at the burden of cardiovascular disease in Israel and its relation to ambient air pollution. Standardized mortality ratios due to cardiovascular disease are significantly elevated in the Haifa Bay Area in comparison to the rest of the country; mortality due to MI is 13% above national average while total ischemic heart disease mortality is 29% above national average. The Haifa Bay Area has a long history of industrialization including possessing the nation's largest oil refineries, oil-fired power plant, agrochemical and cement producers, industrial incinerators and the Eastern Mediterranean's busiest port. The presence of industrial and mobile sources, combined with a basin effect has contributed to air pollution in the Haifa Bay Area and has raised concerns about potential health effects.

Research Hypothesis- Fine particulate variation in the Haifa Bay Area is positively associated with emergency room visit,hospitalization rates and mortality rates secondary to cardiovascular disease.

Study Methodology- Critical to any environmental epidemiology research is coordination between experts in exposure assessment and health outcomes. This study will be a two year collaborative effort between the School of Public Health at the University of Haifa and the Faculty of Civil and Environmental Engineering at the Technion. Exposure measures will come from the Haifa District Municipal Association for the Environment's (HDMAE) network of 15 monitoring stations in the region. HDMAE also monitors a number of meteorological covariates (ie. maximum and minimum temperatures, mean humidity, and mean barometric pressure) which will be incorporated into exposure modeling.

Primary outcomes of interest will be daily mortality rates and daily rates of cardiovascular related emergency room visits and hospitalizations at the Rambam Medical Center in Haifa Israel. Electronic medical record databases will be queried for ICD-9 codes of related cardiac (acute coronary syndrome, heart failure, dysrhythmia/conduction disturbance) diagnoses. A time-series analysis will be utilized to assess change in mortality and emergency room visit rates in relation to incremental change in PM2.5. Covariates in the model will include seasonal trends in disease incidence, daily concentration of co-pollutants, meteorological variables such as temperature and humidity. Calculation of relative risk will incorporate a 1 through 7 day lag into the model into to determine latency of effect.

Contribution to Environmental Health in Israel- This research hopes to evaluate the contribution of ambient air pollution on the increased rate of cardiovascular morbidity in the Haifa Bay Area. In assessing effect modification in sub-groups we will contribute to the understanding of how environmental pollution impacts Israel's diverse population. In calculating the economic impact of associated morbidity and mortality we hope to contribute to the cost-benefit analysis of environmental regulation in Israel. Finally, by creating prediction models of daily cardiovascular emergency department visits based on air pollution and meteorlogical variation, we can potentially inform local medical facilities and public health agencies on how to predict and prepare for changes in disease incidence.

ELIGIBILITY:
Inclusion Criteria:

* All Patients visiting the ER between Jan 2009 and Dec 2010 at the Rambam Medical Center in Haifa Israel.

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients visiting the ER between Jan 2009 and Dec 2010 at the Rambam Medical Center in Haifa Israel. Electronic medical record databases will be queried for ICD-9 codes of related cardiac (acute coronary syndrome, heart failure, dysrhythmia/conduction disturbance) diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-04

CONTACTS AND LOCATIONS:
Overall Officials: Haim Hammerman, prof, Principal Investigator — Rambam Health Care Campus